CLINICAL TRIAL: NCT07394530
Title: A Comparative Study of In Vitro Fertilization Outcomes Between PPOS and Antagonist Protocols in Women With Polycystic Ovary Syndrome
Brief Title: Comparison of IVF Outcomes Between PPOS and Antagonist Protocols in Women With PCOS
Acronym: PPOS-PCOS-IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi General Hospital (Vietnam) (Other)
Responsible Party: Principal Investigator, Nguyen Duy Phuong, Medical Doctor, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGH-IVF-PCOS-PPOS-ANT-2026; HMUIRB2402 (Other: Hanoi Medical University Institutional Review Board); 05/CN-BVĐKHN (Other: Ethics Committee in Biomedical Research, Hanoi Department of Health)
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Female Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPOS Protocol (Experimental): Participants receive ovarian stimulation using the progestin-primed ovarian stimulation (PPOS) protocol for in vitro fertilization.
  Interventions: Drug: Progestin-Primed Ovarian Stimulation (PPOS)
- GnRH Antagonist Protocol (Active Comparator): Participants receive ovarian stimulation using a GnRH antagonist protocol for in vitro fertilization.
  Interventions: Drug: GnRH Antagonist Protocol

INTERVENTIONS:
Drug: Progestin-Primed Ovarian Stimulation (PPOS) — Ovarian stimulation using a progestin-primed ovarian stimulation (PPOS) protocol, including gonadotropins combined with oral progestin for pituitary suppression during in vitro fertilization treatment.
  Arms: PPOS Protocol
Drug: GnRH Antagonist Protocol — Ovarian stimulation using a gonadotropin-releasing hormone (GnRH) antagonist protocol for pituitary suppression during in vitro fertilization treatment.
  Arms: GnRH Antagonist Protocol

SUMMARY:
This study aims to compare the outcomes of two ovarian stimulation protocols used in in vitro fertilization (IVF): the progestin-primed ovarian stimulation (PPOS) protocol and the GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years
* Diagnosed with polycystic ovary syndrome (PCOS) according to the modified Rotterdam criteria (2004) (≥2 of 3: oligo/anovulation, hyperandrogenism, or polycystic ovarian morphology on ultrasound)
* Indicated for in vitro fertilization (IVF) due to PCOS alone or PCOS with other infertility factors (e.g., tubal factor, previous failed IUI)
* Eligible for controlled ovarian stimulation for IVF
* Husband/partner with normal sperm parameters or mild to moderate oligoasthenoteratozoospermia (OAT)
* Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

* Uterine abnormalities that may impair implantation or pregnancy outcomes, including congenital uterine malformations, large fibroids distorting the uterine cavity, adenomyosis, or severe intrauterine pathology.
* History of major ovarian or uterine surgery affecting ovarian reserve or uterine structure (e.g., ovarian cystectomy, endometriosis surgery, myomectomy, unilateral oophorectomy)
* History of recurrent pregnancy loss (≥3 spontaneous miscarriages)
* Known chromosomal abnormalities in either partner
* Inability to adhere to study protocol or follow-up procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants with polycystic ovary syndrome (PCOS) who are indicated for IVF treatment are eligible for this study
Enrollment: 400 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate at 12 weeks | Up to 12 weeks after embryo transfer
  Ongoing pregnancy defined as a viable intrauterine pregnancy with fetal cardiac activity confirmed by ultrasound at or beyond 12 weeks of gestation.

SECONDARY OUTCOMES:
Number of Oocytes Retrieved | From ovarian stimulation start to oocyte retrieval (approximately 10-14 days)
  Total number of oocytes retrieved per ovarian stimulation cycle at the time of oocyte retrieval
Number of Mature (MII) Oocytes | At the time of oocyte retrieval (approximately 10-14 days after stimulation start)
  Number of mature oocytes at the metaphase II (MII) stage identified at the time of oocyte retrieval
Live birth rate | Up to delivery (approximately 9-12 months after embryo transfer)
  Live birth rate of live-born infants at ≥24 weeks of gestation or with birth weight ≥500 g and signs of life after birth.
Clinical pregnancy rate | 6-7 weeks after embryo transfer
  Clinical pregnancy defined as the presence of a gestational sac with fetal cardiac activity confirmed by ultrasound
Fertilization Rate | 16-18 hours after oocyte insemination
  Fertilization rate, defined as the percentage of fertilized oocytes
Number of Usable Embryos | From fertilization to embryo assessment (approximately Day 3 to Day 5 after oocyte retrieval).

CONTACTS AND LOCATIONS:
Overall Officials: Phuong Duy Nguyen, MD, MS, Principal Investigator — Hanoi General Hospital
Locations (1):
- Hanoi General Hospital, Hanoi, Hanoi, Vietnam